CLINICAL TRIAL: NCT00004235
Title: A Phase II Study of Taxotere and Irinotecan (CPT-11) in Patients With Advanced Adenocarcinoma of the Lower Esophagus, Esophagogastric Junction, and Gastric Cardia
Brief Title: Docetaxel and Irinotecan in Treating Patients With Advanced Cancer of the Esophagus or Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9941; CDR0000067479 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-01-28; First posted 2004-03-03 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinotecan + docetaxel (Experimental): Patients receive irinotecan IV over 90 minutes followed by docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.
  Patients achieving a complete response (CR) receive 2 additional courses after CR. Patients experiencing disease progression after a CR and 2 additional courses may be retreated with irinotecan and docetaxel. Dysphagia, anorexia, and swallowing ability are assessed before the first course of treatment and then at each tumor assessment.
  Patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Drug: docetaxel; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: docetaxel
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of combining docetaxel and irinotecan in treating patients who have advanced cancer of the esophagus or stomach.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective tumor response rate in patients with advanced adenocarcinoma of the lower esophagus, esophagogastric junction, and gastric cardia treated with docetaxel and irinotecan. II. Determine time to progression and overall survival of patients treated treated with this regimen. III. Determine the toxic effects of this regimen in these patients. IV. Assess treatment response in these patients by determining the prevalence of dysphagia, anorexia, and swallowing ability at diagnosis and during treatment with this regimen.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed adenocarcinoma of the lower esophagus, esophagogastric junction, or gastric cardia that is considered unresectable and for which no curative therapy exists No other conventional forms of therapy available that would offer a reasonable chance of cure or significant palliation Gastric cardia is defined as no greater than 5 cm from the esophagogastric junction into the stomach Measurable disease At least 1 lesion that can be accurately measured in at least 1 dimension as at least 20 mm No nonmeasurable lesions only, including: Bone lesions Leptomeningeal disease Ascites Pleural/pericardial effusion Inflammatory breast disease Lymphangitis cutis/pulmonis Abdominal masses not confirmed and followed by imaging techniques Cystic lesions No known untreated or treated symptomatic CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST no greater than ULN (less than 2.5 times ULN if alkaline phosphatase no greater than ULN) Alkaline phosphatase no greater than ULN (4 times ULN if AST no greater than ULN) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No New York Heart Association class III or IV heart disease Neurologic: No grade 2 or greater peripheral neuropathy of any etiology No uncontrolled seizure disorder Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Ability to complete questionnaires alone or with assistance No uncontrolled infection No chronic debilitating disease No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or other noninvasive carcinoma

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy or biologic therapy for recurrent or metastatic disease No concurrent biologic therapy No concurrent filgrastim (G-CSF) as primary prophylaxis Chemotherapy: Prior adjuvant chemotherapy after complete resection of original tumor allowed Prior neoadjuvant chemotherapy allowed No prior chemotherapy for recurrent or metastatic disease No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: Prior adjuvant radiotherapy after complete resection of original tumor allowed Prior neoadjuvant radiotherapy allowed At least 4 weeks since prior radiotherapy No prior radiotherapy for recurrent or metastatic disease No prior radiotherapy to more than 25% of bone marrow No concurrent radiotherapy except to CNS Surgery: See Disease Characteristics Prior surgical resection of primary tumor allowed At least 4 weeks since prior abdominal exploration with resection (3 weeks without resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2000-01; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
objective tumor response rate | Up to 5 years

SECONDARY OUTCOMES:
time to progression | Up to 5 years
overall survival | Up to 5 years
treatment response | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Jatoi A, Foster NR, Egner JR, Burch PA, Stella PJ, Rubin J, Dakhil SR, Sargent DJ, Murphy BR, Alberts SR. Older versus younger patients with metastatic adenocarcinoma of the esophagus, gastroesophageal junction, and stomach: a pooled analysis of eight consecutive North Central Cancer Treatment Group (NCCTG) trials. Int J Oncol. 2010 Mar;36(3):601-6. doi: 10.3892/ijo_00000535. PMID 20126980
- [Result] Jatoi A, Tirona MT, Cha SS, Alberts SR, Rowland KM, Morton RF, Nair S, Kardinal CG, Stella PJ, Mailliard JA, Sargen D, Goldberg RM. A phase II trial of docetaxel and CPT-11 in patients with metastatic adenocarcinoma of the esophagus, gastroesophageal junction, and gastric cardia. Int J Gastrointest Cancer. 2002;32(2-3):115-23. doi: 10.1385/ijgc:32:2-3:115. PMID 12794247
- [Result] Tria Tirona M, Jatoi A, Cha SS, et al.: A phase II trial of CPT-11 and docetaxel in patients with metastatic esophageal cancer: preliminary toxicity data from the North Central Cancer Treatment Group. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-605, 2002.